CLINICAL TRIAL: NCT03721029
Title: Can Intraoperative Nerve Monitoring Predict and Improve Functional Outcomes After Robotic-assisted Radical Prostatectomy
Brief Title: Intraoperative Nerve Monitoring During Robotic-assisted Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Alexander Nolsøe, MD, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-6-2013-003
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Humans; Urinary Incontinence; Male Urogenital Diseases; Prostatectomy; Erectile Dysfunction
Keywords: Urinary incontinence; Prostate cancer; Erectile dysfunction; Functional outcome; Robotic prostatectomy; Prostatectomy; Urethral sphincter
MeSH Terms: conditions — Urinary Incontinence; Male Urogenital Diseases; Erectile Dysfunction; Prostatic Neoplasms | interventions — Intraoperative Neurophysiological Monitoring

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intraoperative nerve monitoring (Experimental): Patients that undergo robotic-assisted radical prostatectomy with the use intraoperative nerve monitoring, via electromyography, to identify the exact location of the somatic fibers in the pelvic nerves that seem crucial for urinary continence control and erectile function
  Interventions: Device: Intraoperative nerve monitoring,
- Control Cohort (Active Comparator): Patients that undergo standard of care robotic-assisted radical prostatectomy.
  Interventions: Procedure: standard of care robotic-assisted radical prostatectomy

INTERVENTIONS:
Device: Intraoperative nerve monitoring, — Intraoperative nerve monitoring, via electromyography, enables real-time identification of the location of the somatic fibers in the pelvic nerves that seem crucial for urinary continence control and erectile function.
  Arms: Intraoperative nerve monitoring
Procedure: standard of care robotic-assisted radical prostatectomy — With out the usage of intraoperative nerve monitoring
  Arms: Control Cohort

SUMMARY:
The purpose of this study is to evaluate whether the use of intraoperative nerve monitoring during robotic-assisted radical prostatectomy (RARP) can predict and improve post-surgery urinary continence and erectile function.

DETAILED DESCRIPTION:
Study design:

This is a single center, randomized, single blinded, prospective, clinical trial. The study population will comprise of 100 men that will undergo either a non-nerve sparring or unilateral-nerve sparring RARP. This means that the preoperative evaluation has suggested that it will not be possible to preserve the cavernous parasympathetic nerves lying in the fascia on either side of the prostate gland during surgery (called bilateral-nerve sparring). Despite the term, non-nerve sparring surgery, the surgeon will still attempt to preserve the somatic fibers of the pudendal nerve as best possible. However, due to the extent of cancer tissue the surgeon will generally need to operate closer to the pudendal nerve then when performing bilateral-nerve sparring surgery. So, the somatic fibers of the pudendal nerve are more likely to be severed. The same is the case on one side when performing unilateral surgery.

The treatment group will consist of 50 subjects that will undergo nerve monitoring during RARP. Results will be compared to a control cohort consisting of 50 patients that will undergo contemporary RARP.

Aside from the usage of nerve monitoring in the intervention-group, all procedures and care from admission to the hospital through discharge will be standard of care for subjects in both the control and Intervention-group.

Baseline evaluation and collection of data:

Patients will be screened for eligibility on the phone, and if eligible and they accept they will be scheduled to a visit at the hospital where the following data will be registered for all participants prior to surgery:

* Age at time of surgery
* Known co-morbidity
* Body Mass Index (BMI)
* Medicine status
* Smoking
* Partner status
* Level of education
* Employment Clinical status
* Clinical stage (cT-staging)
* Gleason score
* Prostate specific antigen (PSA)

Prior to surgery participants will also have answered the questionnaires listed either prior to or during the first visit and have undergone an MRI and the bulbocavernosus-reflex test:

* ICIQ (International Consultation on Incontinence Questionnaire) form about incontinence symptoms
* Danish Prostate Symptom Score (DAN-PSS)
* International Prostate Symptom Score (IPSS)
* International Index of Erectile Function (IIEF) score
* Erection Hardness Scale (EHS) score
* Presence or absence of bulbocavernosus-reflex. The physician test for this by shortly squeezing the penis while observing if the urethra retracts or the anal sphincter contracts. The test is not painful and only takes a few seconds.
* Magnetic Resonance Imaging (MRI) scan with measurements of the urethral length and width, and prostate volume along with other specific anatomical structures in relation to the urethra. Contrast agents will not be applied.

Intraoperative data:

* Contraction of the sphincter musculature during stimulation via the nerve monitoring system before removal of the prostate gland
* Contraction of the sphincter musculature during stimulation via the nerve monitoring system after removal of the prostate gland.
* Blood loss
* Non- or unilateral nerve sparring
* Lymph node dissection
* Total surgical time
* Sphincter lesion
* The surgeon's subjective prediction whether the patient will return to continence postoperatively

During the procedure, through discharge and before follow-up regime begins, the following data points will be collected:

* Time to removal of catheter
* Leakage of the anastomosis
* Stricture.
* Other adverse effects
* Pathologic cancer stage (pT-stage)
* Pathologic Gleason score
* Status of surgical margins

Follow-up evaluation.

Subjects will be evaluated 14 days after catheter removal and at standard clinical controls at 3, 6 and 12 months. The following questionnaires are answered at every visit:

* International consultation on Incontinence Questionnaire (ICIQ) for incontinence,
* Danish Prostate Symptom Score (DAN-PSS)
* International Prostate Symptom Score (IPSS)
* International Index of Erectile Function (IIEF) and Erection Hardness Scale (EHS).

During the last 3 visits subjects also answers a fluid intake/output questionnaire and hand in the results of a 24-hour pad test. In addition to the questionnaires the patients will also undergo an MRI and a bulbocavernosus reflex test 12 months postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are planned to undergo either non-nerve or unilateral nerve sparring surgery.
* Patients that deemed able to understand the protocol and to return for all the required post-treatment follow-up visits.

Exclusion Criteria:

* Incontinence prior to surgery
* Diabetes
* Known neurological disease that can affect urinary/erectile function
* Condition with Pacemaker
* Previous pelvic trauma
* Previous pelvic surgery including transurethral resection of the prostate
* Previous pelvic radiation therapy

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Return of continence following robotic-assisted radical prostatectomy | 12 months
  Difference in total International consultation on incontinence questionnaire (ICIQ)-score between the 2 groups after a follow-up of 1 year.
  ICIQ is a self-reported survey and screening tool for incontinence. It consists of 3 questions regarding symptoms in the past 4 week, with an overall 0-21 score, where greater values indicate increased severity. Question 1 scores from 0-5, question 2 scores either 0,2,4 or 6 and question 3 scores from 0-10. Only the total score is evaluated. Furthermore there is 1 self-diagnostic question.

SECONDARY OUTCOMES:
Return of erectile function following robotic-assisted radical prostatectomy | 12 months
  Difference in erection rates and sexual activity between the 2 groups after 12 months. Sexual activity defined as yes to the question "Within the last 3 months, have you been sexually active and attempted intercourse?" Erection is defined as a score of at least 17 on the IIEF-5 form and or a score of a least 3 on the EHS form with the use of either no assistance phosphodiesterase 5 inhibitors
Nerve function prior to removal of the prostate correlated to patient's preoperative urinary function | 1 day
  Correlation between nerve signal prior to removal of the prostate and preoperative urinary function
Nerve function prior to removal of the prostate correlated to patient's preoperative erectile function | 1 day
  Correlation between nerve signal prior to removal of the prostate and preoperative erectile function
Nerve function after removal of the prostate correlated to patient's postoperative urinary function | 12 months
  Correlation between nerve signal after removal of the prostate and postoperative urinary function
Nerve function after removal of the prostate correlated to patient's postoperative erectile function | 12 months
  Correlation between nerve signal after removal of the prostate and postoperative erectile function
Difference in the degree of incontinence between the two groups for incontinent patients. | 12 months
  Measured in gram on the 24-hour pad test
Difference in Time to continence between the two groups | 12 months
  Difference in Time to continence between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Jens Sønksen, Dr., Phd, MD, Study Director — Professor
Locations (1):
- Herlev and Gentofte Hospital, Herlev, Central Region, Denmark